CLINICAL TRIAL: NCT06407752
Title: Anthropometric Parameters, Physical Fitness and Muscle Strength in School Going Children
Brief Title: Anthropometric Characteristics, Level of Physical Fitness, and Muscle Strength in Youngsters Attending School
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS/23/0782
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Child Rearing
Keywords: Anthropometric parameter; Dynamometer; Conicity index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It has long been believed that evaluating a child's development is essential to determining population health trends and creating effective interventions. Assessing school-age children's overall health and well-being in the 7-14 age range requires careful observation of their anthropometric metrics, physical fitness, and muscle strength. These assessments can provide insight into several physical health-related concerns during this crucial period of childhood development. Anthropometric parameters include height (in centimeters or centimeters), body mass index (BMI), skin fold measurements (which provide estimates of body fat), circumference measurements, and body weight (kg), which is typically measured in kilograms (kg).

A cross-sectional descriptive study design will be used. The goal of this research is to determine how anthropometric characteristics, physical

DETAILED DESCRIPTION:
The participants' anthropometric parameters will be assessed both subjectively and objectively to calculate the data. Weight will be measured in kilograms using a weight machine, and height will be measured in inches using a measuring tape and converted into meters, respectively, to determine BMI. Using a measuring tape, the chest, abdomen, thigh, triceps, and supraillium are measured to determine the skin fold measurement, which determines the body fat percentage. Circumference measurements, such as those taken of the midthigh, biceps, waist, hips, and conicity index. The body mass index, conicity index, weight scale, and inch tape will be used for these measurements.

A common tool is the International Physical Activity Questionnaire (IPAQ). The seven-day IPAQ-SF is a self-administered, scientifically validated recall questionnaire for children ages 7 to 14. The quantity of time a child spends exercising during the

ELIGIBILITY:
Inclusion Criteria:

* The age of participants will be 7-14 years.
* Males and females will be included.
* Healthy and physically fit participants will be taken.
* Regular and enrolled students of public and private schools.

Exclusion Criteria:

* Students with any significant past medical or surgical history will be not included in this study.
* Chronic disease or injury to the lower extremity or were on continuous medication

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants will range in age from 7 to 14. Both men and women will be present. Only physically well and in good health will be accepted. Enrolled and regular pupils in both public and private schools.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 8 weeks
  manual muscle testing

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Yousaf, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karim A, Qaisar R. Anthropometric measurements of school-going-girls of the Punjab, Pakistan. BMC Pediatr. 2020 May 16;20(1):223. doi: 10.1186/s12887-020-02135-4. PMID 32416717